CLINICAL TRIAL: NCT01624662
Title: A 16-Week Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study Evaluating the Efficacy and Safety of Intranasal Administration of 100, 200, and 400 μg of Fluticasone Propionate Twice a Day (Bid) Using a Novel Bi-directional Device in Subjects With Bilateral Nasal Polyposis Followed by an 8-week, Open-label Extension Phase to Assess Safety
Brief Title: Efficacy and Safety Study of Intranasal Administration of 100, 200, and 400 μg of Fluticasone Propionate Using a Novel Bi-directional Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-NP-3102
Record Dates: First submitted 2012-06-13; First posted 2012-06-21 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-01

CONDITIONS: Bilateral Nasal Polyposis
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- OPN-375 100 mcg (Active Comparator): Double-Blind Treatment Phase: OPN-375 100 mcg BID x 16 weeks; Open-Label Extension Phase: OPN-375 400 mcg BID x 8 weeks
  Interventions: Drug: Fluticasone propionate
- OPN-375 200 mcg (Active Comparator): Double-Blind Treatment Phase: OPN-375 200 mcg BID x 16 weeks; Open-Label Extension Phase: OPN-375 400 mcg BID x 8 weeks
  Interventions: Drug: Fluticasone propionate
- OPN-375 400 mcg (Active Comparator): Double-Blind Treatment Phase: OPN-375 400 mcg BID x 16 weeks; Open-Label Extension Phase: OPN-375 400 mcg BID x 8 weeks
  Interventions: Drug: Fluticasone propionate
- Placebo (Placebo Comparator): Double-Blind Treatment Phase: Matched Placebo BID x 16 weeks; Open-Label Extension Phase: OPN-375 400 mcg BID x 8 weeks
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone propionate — Delivered via Optinose Exhalation Delivery System
  Other Names: OPN-375

SUMMARY:
The primary objective of this study was to compare the efficacy of intranasal administration of 100, 200, and 400 μg twice daily (bid) of fluticasone propionate, delivered by the Optinose device, with matching placebo in subjects with bilateral nasal polyposis and nasal congestion.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel-group, multicenter study designed to assess the efficacy and safety of intranasal administration of 3 doses of fluticasone propionate (100, 200, and 400 μg bid), delivered by the Optinose device, in subjects with bilateral nasal polyposis and nasal congestion.

This study consisted of 3 phases. After signing informed consent, subjects who met eligibility criteria at Visit 1 (screening) visit entered the study.

1. Pretreatment phase (single-blind, placebo, run-in): 7 to 14 days duration, to determine disease status eligibility and to ensure the subject was able to comply with study procedures prior to randomization and enrolment in the double-blind treatment phase
2. Double-blind treatment phase: 16 weeks duration with 6 scheduled visits starting with Visit 2 (Day 1) when eligible subjects were randomized by balance allocation to 1 of 4 treatment groups and ending at Visit 7 (Week 16)
3. Open-label extension phase: 8 weeks duration with 1 scheduled visit (Visit 8 [Week 24]), during which all subjects received fluticasone propionate 400 mcg BID delivered by the Optinose device

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older
* Women must

  * be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
  * be surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation at least 1 year before screening) or otherwise be incapable of pregnancy, or
  * be postmenopausal (spontaneous amenorrhea for at least 1 year).
* Women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (B-hCG) or urine pregnancy test (depending on local regulations) at the screening visit
* Must have bilateral nasal polyposis with a grade of 1 to 3 in each of the nasal cavities as determined by the Lildholdt scale score measured by nasoendoscopy at both screening and baseline visits
* Must have at least moderate symptoms of nasal congestion/obstruction as reported by the subject for the 7 day period preceding the screening visit
* At the baseline visit (Day 1), must have a morning score of at least 2 (moderate) on nasal congestion/obstruction recorded on the subject diary for at least 5 of the last 7 days of the 7 to up to 14 day run-in period
* Must demonstrate an ability to correctly complete the daily diary during the run-in period to be eligible for randomization
* Subjects with comorbid asthma or COPD must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use) within the 3 months before the screening visit. Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent) for at least 3 months before screening with plans to continue use throughout the study.
* Must be able to cease treatment with intranasal medications including, but not limited to, intranasal steroids, intranasal sodium cromolyn, nasal atropine, nasal ipratropium bromide, inhaled corticosteroids (except permitted doses listed above for comorbid asthma and COPD) at the screening visit
* Must be able to cease treatment with oral and nasal decongestants and antihistamines at the screening visit
* Must be able to use the OptiNose device correctly; all subjects will be required to demonstrate correct use of the placebo device at screening, Visit 1.
* Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Women who are pregnant or lactating
* Have complete or near-complete obstruction of the nasal cavities
* Inability to achieve bilateral nasal airflow for any reason including nasal septum deviation
* Inability to have each nasal cavity examined for any reason including nasal septum deviation
* Nasal septum perforation
* Has had more than 1 episode of epistaxis with frank bleeding in the month before the screening visit
* Have evidence of significant baseline mucosal injury, ulceration or erosion (eg, exposed cartilage, perforation) on baseline nasal examination/nasal endoscopy
* History of more than 5 sinonasal surgeries for either nasal polyps or nasal/sinus inflammation (lifetime)
* History of sinus or nasal surgery within 6 months before the screening visit
* History of any surgical procedure that prevents the ability to accurately grade polyps
* Have symptoms of seasonal allergic rhinitis at screening or baseline and/or, based on time of year, would anticipate onset of symptoms within 4 weeks of randomization
* Current, ongoing rhinitis medicamentosa (rebound rhinitis)
* Have significant oral structural abnormalities, eg, a cleft palate
* Diagnosis of cystic fibrosis
* History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
* Purulent nasal infection, acute sinusitis, or upper respiratory tract infection within 2 weeks before the screening visit. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution Note: Subjects who are taking prophylactic antibiotics will be allowed to enter the study as long as they intend to continue the antibiotics for the duration of the study.
* Planned sinonasal surgery during the period of the study
* Allergy, hypersensitivity, or contraindication to corticosteroids or steroids
* Allergy or hypersensitivity to any excipients in study drug
* Exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before the screening visit; except as noted in inclusion criteria for subjects with comorbid asthma or COPD
* Have nasal candidiasis
* Have taken a potent CYP3A4 inhibitor within 14 days before the screening visit.
* History or current diagnosis of any form of glaucoma or ocular hypertension (ie, >21 mmHg)
* History of intraocular pressure elevation on any form of steroid therapy
* History or current diagnosis of the presence (in either eye) of a cataract
* Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
* A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol use, abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
* Positive urine drug screen at screening visit for drugs of abuse, with the exception of prescribed medications for legitimate medical conditions
* Have participated in an investigational drug clinical trial within 30 days of the screening visit
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2015-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Bensch Clinical Research LLC, Stockton, California
  - Colorado Allergy & Asthma Centers, PC, Centennial, Colorado
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - University of Vermont, Burlington, Vermont
  - Bellingham Asthma, Allergy, and Immunology Clinic, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: Yes
randomization codes sent to PIs

REFERENCES:
- [Derived] Ow RA, McGinnis JP 2nd, Sacks HJ, Mehle ME. The Effect of EDS-FLU on Objective and Patient-Reported Subjective Outcomes for Patients with Chronic Rhinosinusitis with Nasal Polyps. Ear Nose Throat J. 2025 Feb;104(2):93-101. doi: 10.1177/01455613221088698. Epub 2022 Apr 18. PMID 35437059
- [Derived] Skoner DP, Meltzer EO, Skoner J, Sacks HJ, Lumry WR. Evaluation of the ocular safety associated with the exhalation delivery system with fluticasone. Allergy Asthma Proc. 2022 Jan 9;43(1):70-77. doi: 10.2500/aap.2022.43.210096. Epub 2021 Nov 9. PMID 34753535
- [Derived] Leopold DA, Elkayam D, Messina JC, Kosik-Gonzalez C, Djupesland PG, Mahmoud RA. NAVIGATE II: Randomized, double-blind trial of the exhalation delivery system with fluticasone for nasal polyposis. J Allergy Clin Immunol. 2019 Jan;143(1):126-134.e5. doi: 10.1016/j.jaci.2018.06.010. Epub 2018 Jun 19. PMID 29928924

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matched placebo BID x 16 weeks, then OPN-375 400 mcg BID (open-label) x 8 weeks
- OPN-375 100 mcg: OPN-375 100 mcg BID x 16 weeks, then OPN-375 400 mcg BID (open-label) x 8 weeks
- OPN-375 200 mcg: OPN-375 200 mcg BID x 16 weeks, then OPN-375 400 mcg BID (open-label) x 8 weeks
- OPN-375 400 mcg: OPN-375 400 mcg BID x 16 weeks, then OPN-375 400 mcg BID (open-label) x 8 weeks
Period: Double-Blind Treatment Phase (Wks 1-16)
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Started | 80 | 81 | 80 | 82
Completed | 70 | 78 | 76 | 82
Not Completed | 10 | 3 | 4 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 5 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 0
Period: Open-Label Extension Phase (Wks 17-24)
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Started | 70 | 78 | 72 | 79
Completed | 69 | 76 | 71 | 78
Not Completed | 1 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matched placebo BID x 16 weeks, then OPN-375 400 mcg BID x 8 weeks
- OPN-375 100 mcg: OPN-375 100 mcg BID x 16 weeks, then OPN-375 400 mcg BID x 8 weeks
- OPN-375 200 mcg: OPN-375 200 mcg BID x 16 weeks, then OPN-375 400 mcg BID x 8 weeks
- OPN-375 400 mcg: OPN-375 400 mcg BID x 16 weeks, then OPN-375 400 mcg BID x 8 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg | Total
Number analyzed (Participants) | 80 | 81 | 80 | 82 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.95) | 46.7 (13.72) | 44.8 (12.87) | 45.0 (12.14) | 45.8 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 34 | 26 | 137
  Male | 42 | 42 | 46 | 56 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76 | 76 | 76 | 76 | 304
  Black or African American | 3 | 3 | 3 | 4 | 13
  Asian | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 1 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 9 | 39
  Poland | 31 | 34 | 33 | 33 | 131
  Romania | 15 | 13 | 13 | 14 | 55
  Ukraine | 12 | 14 | 13 | 15 | 54
  South Africa | 12 | 10 | 11 | 11 | 44
Total Polyp Grading Score (sum of scores from both nasal cavities) [Mean (Standard Deviation); unit: units on a scale] — Nasal Polyp Grading Score (sum of scores from both nasal cavities measured by nasoendoscopy)
  0: No polyps
  1. Mild polyposis - polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis - polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis - large polyps reaching below the lower inferior border of the inferior turbinate Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 3.8 (1.08) | 3.8 (0.98) | 3.9 (1.05) | 3.9 (0.98) | 3.8 (1.02)
Use of ICS treatment for polyps in past 10 years [Count of Participants; unit: Participants] | 73 | 67 | 70 | 70 | 280
Previous sinus surgery for polyp removal or sinus surgery [Count of Participants; unit: Participants] — Subjects may have had both sinus surgery and polypectomy.
  Participants | 24 | 28 | 33 | 26 | 111
Previous polyp removal surgery via polypectomy only [Count of Participants; unit: Participants] — Subjects may have had both sinus surgery and polypectomy.
  Participants | 30 | 33 | 25 | 27 | 115
Nasal Congestion/obstruction Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects used an electronic diary to record nasal symptoms each morning for the 7-day period preceding the screening visit, evaluating symptom severity immediately preceding the time of scoring (instantaneous).
  Nasal Symptom Score
  0: None
  1. Mild - symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - definite awareness of symptoms that is bothersome but tolerable
  3. Severe - symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 2.29 [1.6 to 3.0] | 2.23 [1.6 to 3.0] | 2.20 [1.7 to 3.0] | 2.25 [1.6 to 3.0] | 2.24 [1.6 to 3.0]
Rhinorrhea Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects used an electronic diary to record nasal symptoms each morning for the 7-day period preceding the screening visit, evaluating symptom severity immediately preceding the time of scoring (instantaneous).
  Nasal Symptom Score
  0: None
  1. Mild - symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - definite awareness of symptoms that is bothersome but tolerable
  3. Severe - symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 1.8 [0.0 to 3.0] | 1.89 [0.0 to 3.0] | 1.86 [0.0 to 3.0] | 1.77 [0.0 to 3.0] | 1.83 [0.0 to 3.0]
Facial Pain or Pressure Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects used an electronic diary to record nasal symptoms each morning for the 7-day period preceding the screening visit, evaluating symptom severity immediately preceding the time of scoring (instantaneous).
  Nasal Symptom Score
  0: None
  1. Mild - symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate - definite awareness of symptoms that is bothersome but tolerable
  3. Severe - symptoms that are hard to tolerate, cause interference with activities or daily living Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 1.46 [0.0 to 3.0] | 1.46 [0.0 to 3.0] | 1.48 [0.0 to 3.0] | 1.35 [0.0 to 3.0] | 1.44 [0.0 to 3.0]
Hyposmia Score (7-day instantaneous morning) [Mean (Full Range); unit: units on a scale] — Subjects used an electronic diary to record nasal symptoms each morning for the 7-day period preceding the screening visit, evaluating symptom severity immediately preceding the time of scoring (instantaneous).
  Hyposmia Score
  0: Normal
  1. Slightly impaired
  2. Moderately impaired
  3. Absent Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 2.47 [0.0 to 3.0] | 2.36 [0.0 to 3.0] | 2.54 [0.9 to 3.0] | 2.33 [0.0 to 3.0] | 2.43 [0.0 to 3.0]
Sinonasal Outcome Test 22 (SNOT-22) Total Score [Mean (Full Range); unit: units on a scale] — SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as it can be Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 52.0 [14 to 94] | 48.5 [9 to 97] | 48.1 [11 to 92] | 47.1 [7 to 103] | 48.9 [7 to 103]
Medical Outcomes Study Sleep Scale Revised (MOS Sleep-R) [Mean (Full Range); unit: units on a scale] — The MOS Sleep-R is a brief, self-administered, validated questionnaire designed to measure key aspects of sleep, such as disturbance, adequacy, somnolence, and quantity. The 12-item version with a 4-week recall was used in this study. The score range for the 12-item version is 0 to 100, lower scores indicating better sleep and higher scores indicating worse sleep. The scale yields a Sleep Problem Index and scores on the following 6 subscales: Sleep Disturbance, Snoring, Shortness of Breath or Headache, Sleep Adequacy, Sleep Somnolence, and Sleep Quantity. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 41.7 [5.6 to 86.1] | 40.9 [8.3 to 94.4] | 43.0 [2.8 to 86.1] | 39.1 [0.0 to 77.8] | 41.2 [0.0 to 94.4]
Rhinosinusitis Disability Index (RSDI) Total Score [Mean (Full Range); unit: units on a scale] — The RSDI is a subject-completed instrument that evaluates the self-perceived impact of disease specific head and neck disorders. The RSDI has 30 items in 3 domains: Physical (11 items), Functional (9 items), and Emotional (10 items). The RSDI scale ranges from 0-120, 0 being better quality of life and less impact of CRS on daily function and 120 being worse quality of life and more impact of CRS on daily function. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 44.9 [4 to 98] | 43.9 [7 to 111] | 39.7 [2 to 89] | 41.5 [0 to 85] | 42.5 [0 to 111]
Short Form (36) Health Survey Version 2 (SF-36v2) - Mental Component [Mean (Full Range); unit: units on a scale] — The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 43.1 [21.5 to 63.58] | 44.4 [12.27 to 61.03] | 45.9 [19.63 to 64.81] | 47.0 [20.6 to 61.63] | 45.1 [12.27 to 64.81]
Short Form (36) Health Survey Version 2 (SF-36v2) - Physical Component [Mean (Full Range); unit: units on a scale] — The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health perceptions. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  units on a scale
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 45.8 [26.97 to 60.07] | 46.1 [28.61 to 58.86] | 46.5 [29.56 to 59.43] | 46.4 [22.64 to 60.32] | 46.2 [22.64 to 60.32]
Peak Nasal Inspiratory Flow (PNIF) [Mean (Full Range); unit: L/min] — The PNIF is an assessment of nasal passage obstruction and was measured using an In-Check portable nasal inspiratory flow meter. To measure PNIF, a mask was placed over the nose during inspiration and inspiratory flow was recorded. Each subject inhaled 3 times and each measurement was recorded. The PNIF value used was the greatest of the 3 results at each time point. Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  L/min
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 119.7 [30 to 370] | 123.4 [30 to 370] | 107.6 [40 to 350] | 122.7 [30 to 370] | 118.4 [30 to 370]
Nasal Polyp Surgery Eligibility [Count of Participants; unit: Participants] — A subject was considered eligible for surgical intervention if the following conditions were met:
  * Subject has had moderate symptoms of congestion from nasal polyposis for ≥ 3 months.
  * Subject continues to suffer from at least moderate symptoms despite use of topical steroids at conventional doses for ≥ 6 weeks.
  * Subject continues to suffer from at least moderate symptoms despite use (or previous use) of saline lavage for ≥ 6 weeks.
  * Subject has endoscopically visualized bilateral nasal polyposis of at least moderate severity (nasal polyp grading score ≥ 2 in at least 1 nostril). Population: These data are reported for the Full Analysis Set, which included all subjects who received at least one dose of study drug, and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
  Participants
    number analyzed (Participants) | 79 | 80 | 80 | 82 | 321
    (all) | 45 | 40 | 42 | 45 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change in 7-day Average Instantaneous Morning Diary Congestion/Obstruction Symptoms
Description: Subjects reported nasal symptoms using the electronic diary twice daily immediately before dosing.
  0: None
  1. Mild, symptoms clearly present, but minimal awareness, and easily tolerated
  2. Moderate, definite awareness of symptoms that is bothersome but tolerable
  3. Severe, symptoms that are hard to tolerate, cause interference with activities or daily living
  During the single-blind run-in phase and during the 16-week, double-blind treatment phase, an electronic diary was provided to each subject. Subjects reported both instantaneous (evaluation of symptom severity immediately preceding the time of scoring) and reflective (evaluation of symptoms severity over the previous 12 hours) scores for nasal congestion/obstruction symptoms.
Time Frame: Baseline, Week 4 of the double-blind treatment phase
Population: The Full Analysis Set includes subjects who received at least one dose of study drug and who had baseline assessments of polyp size (nasoendoscopy) and recorded morning nasal congestion/obstruction symptoms.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Matched placebo BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
- OPN-375 100 mcg: OPN-375 100 mcg BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
- OPN-375 200 mcg: OPN-375 200 mcg BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
- OPN-375 400 mcg: OPN-375 400 mcg BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 79 | 80 | 80 | 82
units on a scale | -0.24 (0.07) | -0.59 (0.07) | -0.68 (0.07) | -0.62 (0.07)

2. Primary Outcome: Change in Total Polyp Grade
Description: Determined by a nasal polyp grading scale score (sum of scores from both nasal cavities) measured by nasoendoscopy
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 79 | 80 | 80 | 82
units on a scale | -0.61 (0.11) | -1.31 (0.11) | -1.22 (0.11) | -1.41 (0.10)

3. Secondary Outcome: Nasal Congestion/Obstruction Score (7-day Instantaneous Morning)
Description: Measured by the 7-day average instantaneous morning diary symptom scores
Time Frame: Week 16 of the double-blind treatment phase
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 69 | 77
units on a scale | -0.48 (0.09) | -0.99 (0.09) | -0.93 (0.09) | -0.97 (0.09)

4. Secondary Outcome: Change in Rhinorrhea Score (7-day Instantaneous Morning)
Description: Change from baseline in rhinorrhea symptoms, as measured by AM and PM diary symptom scores
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Population: Missing data were imputed using the multiple imputation method in the primary analyses for the co-primary efficacy variables. For other efficacy analyses, missing or invalid values were not imputed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 69 | 77
units on a scale | -0.42 (0.09) | -1.00 (0.09) | -0.84 (0.09) | -0.84 (0.08)

5. Secondary Outcome: Facial Pain or Pressure Score (7-day Instantaneous Morning)
Description: Change from baseline in facial pain/pressure symptoms, as measured by AM and PM diary symptom scores
Time Frame: Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 69 | 77
units on a scale | -0.48 (0.09) | -0.85 (0.09) | -0.81 (0.09) | -0.75 (0.08)

6. Secondary Outcome: Hyposmia Score (7-day Instantaneous Morning)
Description: Change from baseline in hyposmia symptoms, as measured by AM and PM diary symptom scores
Time Frame: Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 69 | 77
units on a scale | -0.24 (0.10) | -0.54 (0.09) | -0.47 (0.10) | -0.63 (0.09)

7. Secondary Outcome: Change in Total Nasal Polyp Score
Description: Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
  Determined by a nasal polyp grading scale score (sum of scores from both nasal cavities measured by nasoendoscopy)
Time Frame: Baseline, Week 24 of the open-label extension phase
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 69 | 78
units on a scale | -1.06 (0.12) | -1.60 (0.11) | -1.48 (0.12) | -1.75 (0.11)

8. Secondary Outcome: Polyp Grade of 0 in at Least One Nostril
Description: Subjects with a Polyp Grade of 0 (None) in at least one nostril
  Polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy. This outcome measured how many patients with a polyp grad of 0 in at least 1 nostril.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior border of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis large polyps reaching below the lower inferior border of the inferior turbinate
Time Frame: Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: Number of patients analyzed at Week 24 is lower as some patients elected not to participate in the open-label extension phase or withdrew during the open-label extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 79 | 73 | 81
Participants
  Week 16 | 3 | 10 | 6 | 11
  Week 24 (all pts on OPN-375 400 μg BID wks 17-24): number analyzed (Participants) | 69 | 77 | 69 | 78
  Week 24 (all pts on OPN-375 400 μg BID wks 17-24) | 6 | 19 | 17 | 22

9. Secondary Outcome: Sinonasal Outcome Test 22 (SNOT-22) Total Score
Description: SNOT-22 is a subject-completed questionnaire that consists of 22 questions. The questions on the SNOT-22 efficacy evaluation were used to calculate a total score. 22 questions are divided among 4 subscales: Rhinologic (7 questions), Ear/Facial Symptoms (4 questions), Sleep Function (3 questions), and Psychological Issues (6 questions). Each item was rated on the 5-point scale. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as it can be
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 68 | 79 | 74 | 81
units on a scale
  Week 16 | -11.70 (1.81) | -21.14 (1.71) | -21.43 (1.75) | -21.05 (1.68)
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 67 | 76 | 69 | 78
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | -19.45 (1.85) | -22.89 (1.75) | -22.92 (1.80) | -23.21 (1.72)

10. Secondary Outcome: MOS Sleep-R Score
Description: The MOS Sleep-R is a brief, self-administered, validated questionnaire designed to measure key aspects of sleep, such as disturbance, adequacy, somnolence, and quantity. The 12-item version with a 4-week recall was used in this study. The score range for the 12-item version is 0 to 100, lower scores indicating better sleep and higher scores indicating worse sleep. The scale yields a Sleep Problem Index and scores on the following 6 subscales: Sleep Disturbance, Snoring, Shortness of Breath or Headache, Sleep Adequacy, Sleep Somnolence, and Sleep Quantity.
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- OPN 375 200 mcg: OPN-375 200 mcg BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
- OPN 375 400 mcg: OPN-375 400 mcg BID x 16 weeks, then OPN-375 400 mcg (open-label) BID x 8 weeks
Arm/Group | Placebo | OPN-375 100 mcg | OPN 375 200 mcg | OPN 375 400 mcg
Number analyzed (Participants) | 69 | 79 | 74 | 81
units on a scale | -10.03 (1.52) | -14.26 (1.46) | -15.78 (1.50) | -14.30 (1.44)

11. Secondary Outcome: Rhinosinusitis Disability Index (RSDI) Total Score
Description: The RSDI is a subject-completed instrument that evaluates the self-perceived impact of disease specific head and neck disorders. The RSDI has 30 items in 3 domains: Physical (11 items), Functional (9 items), and Emotional (10 items). The RSDI scale ranges from 0-120, 0 being better quality of life and less impact of CRS on daily function and 120 being worse quality of life and more impact of CRS on daily function.
Time Frame: Baseline, Week 16 of the double-blind treatment phase
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 76 | 74 | 81
units on a scale | -7.80 (1.97) | -15.54 (1.86) | -15.37 (1.89) | -16.69 (1.80)

12. Secondary Outcome: SF-36v2 - Mental Component
Description: The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 77 | 74 | 81
units on a scale
  Week 16 | 1.69 (0.86) | 4.37 (0.81) | 3.88 (0.83) | 3.98 (0.80)
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 69 | 74 | 69 | 77
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | 4.90 (0.93) | 4.07 (0.89) | 4.41 (0.92) | 5.86 (0.87)

13. Secondary Outcome: SF-36v2 - Physical Component
Description: The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire that measures 8 domains of health: limitations in physical activities, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, limitations in usual role activities, vitality, and general health perceptions. It yields scale scores for each of the 8 health domains, and 2 summary measures of physical and mental health. Each scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: Baseline, Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 77 | 74 | 81
units on a scale
  Week 16 | 2.78 (0.70) | 4.27 (0.66) | 4.57 (0.67) | 5.07 (0.64)
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 69 | 74 | 69 | 77
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | 5.50 (0.67) | 5.23 (0.64) | 5.85 (0.67) | 6.06 (0.63)

14. Secondary Outcome: Number of Participants in Each Category of PGIC
Description: Patient Global Impression of Change; subject responses to the question: "Since starting the study drug, how would you rate the change in your symptoms?" Percentage includes patients who scored either "very much improved," "much improved," or "minimally improved."
Time Frame: Week 16 of the double-blind treatment phase, Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matched placebo BID x 16 weeks
- 100 mcg Fluticasone Proprionate: 100 mcg fluticasone propionate BID x 16 weeks
- 200 mcg Fluticasone Proprionate: 200 mcg fluticasone propionate BID x 16 weeks
- 400 mcg Fluticasone Prioprionate: 400 mcg fluticasone propionate BID x 16 weeks
Arm/Group | Placebo | 100 mcg Fluticasone Proprionate | 200 mcg Fluticasone Proprionate | 400 mcg Fluticasone Prioprionate
Number analyzed (Participants) | 70 | 78 | 75 | 81
Participants
  Week 16: Very much improved | 6 | 19 | 17 | 24
  Week 16: Much improved | 16 | 34 | 34 | 31
  Week 16: Minimally improved | 22 | 15 | 16 | 19
  Week 16: No change | 18 | 7 | 7 | 7
  Week 16: Minimally worse | 5 | 1 | 0 | 0
  Week 16: Much worse | 2 | 1 | 1 | 0
  Week 16: Very much worse | 1 | 1 | 0 | 0
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 69 | 76 | 69 | 78
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Very much improved | 17 | 21 | 23 | 25
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Much improved | 26 | 37 | 24 | 40
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Minimally improved | 19 | 13 | 15 | 6
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): No change | 3 | 3 | 4 | 6
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Minimally worse | 3 | 1 | 3 | 0
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Much worse | 1 | 1 | 0 | 1
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): Very much worse | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants Eligible for Nasal Polyp Surgery
Description: A subject was considered eligible for surgical intervention if the following conditions were met:
  * Subject has had moderate symptoms of congestion from nasal polyposis for ≥ 3 months.
  * Subject continues to suffer from at least moderate symptoms despite use of topical steroids at conventional doses for ≥ 6 weeks.
  * Subject continues to suffer from at least moderate symptoms despite use (or previous use) of saline lavage for ≥ 6 weeks.
  * Subject has endoscopically visualized bilateral nasal polyposis of at least moderate severity (nasal polyp grading score ≥ 2 in at least 1 nostril).
Time Frame: Week 16 of the double-blind treatment phase; Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 69 | 78 | 73 | 81
Participants
  Week 16 | 23 | 13 | 13 | 17
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 69 | 76 | 69 | 78
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | 13 | 9 | 12 | 11

16. Secondary Outcome: Peak Nasal Inspiratory Flow (PNIF)
Description: The PNIF is an assessment of nasal passage obstruction and was measured using an In-Check portable nasal inspiratory flow meter. To measure PNIF, a mask was placed over the nose during inspiration and inspiratory flow was recorded. Each subject inhaled 3 times and each measurement was recorded. The PNIF value used was the greatest of the 3 results at each time point.
  Change from baseline in Peak Nasal Inspiratory Flow (PNIF)
Time Frame: Week 16 of the double-blind treatment phase; Week 24 of the open-label extension phase
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | OPN-375 100 mcg | OPN-375 200 mcg | OPN-375 400 mcg
Number analyzed (Participants) | 67 | 79 | 74 | 81
L/min
  Week 16 | 0.54 (5.37) | 26.50 (5.12) | 24.92 (5.25) | 28.64 (5.04)
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24): number analyzed (Participants) | 67 | 76 | 69 | 78
  Week 24 (all pts on OPN-375 400 mcg BID wks 17-24) | 15.34 (5.42) | 32.06 (5.20) | 31.87 (5.36) | 33.08 (5.13)

ADVERSE EVENTS:
Groups:
- Placebo (Double-blind Phase): Matched placebo BID x 16 weeks
- OPN-375 100 mcg (Double-blind Phase): OPN-375 100 mcg BID x 16 weeks
- OPN-375 200 mcg (Double-blind Phase): OPN-375 200 mcg BID x 16 weeks
- OPN-375 400 mcg (Double-blind Phase): OPN-375 400 mcg BID x 16 weeks
- OPN-375 400 mcg (Open-label Phase): OPN-375 400 mcg (open-label) BID x 8 weeks
Arm/Group | Placebo (Double-blind Phase) | OPN-375 100 mcg (Double-blind Phase) | OPN-375 200 mcg (Double-blind Phase) | OPN-375 400 mcg (Double-blind Phase) | OPN-375 400 mcg (Open-label Phase)
Serious Adverse Events (participants affected / at risk) | 1/79 | 0/80 | 0/80 | 1/82 | 0/299
Other Adverse Events (participants affected / at risk) | 38/79 | 39/80 | 39/80 | 46/82 | 60/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=79) | OPN-375 100 mcg (Double-blind Phase) (N=80) | OPN-375 200 mcg (Double-blind Phase) (N=80) | OPN-375 400 mcg (Double-blind Phase) (N=82) | OPN-375 400 mcg (Open-label Phase) (N=299)
Meningitis and Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Positional vertigo (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=79) | OPN-375 100 mcg (Double-blind Phase) (N=80) | OPN-375 200 mcg (Double-blind Phase) (N=80) | OPN-375 400 mcg (Double-blind Phase) (N=82) | OPN-375 400 mcg (Open-label Phase) (N=299)
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 3
Bronchitis (Infections and infestations) | 2 | 2 | 2 | 1 | 3
Influenza (Infections and infestations) | 2 | 1 | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1 | 8 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 1 | 2 | 0
URTI (Infections and infestations) | 10 | 4 | 6 | 4 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 3 | 1 | 4
Headache (Nervous system disorders) | 3 | 5 | 6 | 6 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 0
Epistaxis (identified by investigator on routine nasal endoscopy) (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 7 | 8 | 17
Epistaxis (spontaneously reported by subject) (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 12 | 10 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 3 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 8 | 5 | 6
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4 | 4 | 4
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6 | 8 | 9
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes